CLINICAL TRIAL: NCT00668369
Title: Effect of Immunosuppression Drug Weaning on Hepatitis C Virus Induced Liver Damage After Liver Transplantation.
Brief Title: Effect of Immunosuppression Drug Weaning on Hepatitis C Virus (HCV)-Induced Liver Damage After Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Alberto Sanchez-Fueyo, Director IDIBAPS Transplant Immunology Laboratory, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Weaning_HCV
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C Virus Infection; Liver Transplantation
Keywords: Liver Transplantation; Tolerance; Hepatitis C virus infection; Immune responses; Allograft tolerance; Immunosuppression weaning; Immunosuppression minimization
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Liver transplant recipients with HCV infection fulfilling inclusion criteria.
  Interventions: Procedure: Gradual immunosuppression drug withdrawal.

INTERVENTIONS:
Procedure: Gradual immunosuppression drug withdrawal. — Ater obtention of biological samples (peripheral blood, liver tissue) enrolled patients undergo gradual decrease in the doses of immunosuppression drugs (tacrolimus, cyclosporine A and/or mofetil mycophenolate) until complete discontinuation or appearance of rejection.

SUMMARY:
Viral infections can profoundly influence alloimmune responses and hamper allograft tolerance induction. Persistent hepatitis C virus (HCV) infection occurs in 50% of liver and 20% of kidney transplant recipients, but the impact of HCV on the acquisition of allograft tolerance has not been elucidated. Liver transplantation constitutes a unique clinical model to address this question, given that up to 20% of liver recipients can completely discontinue immunosuppressive drugs and attain operational tolerance.

The goal of our study is to determine the influence of HCV-driven immune responses on the acquisition of operational tolerance in liver transplant recipients following drug weaning, and to assess whether immunosuppression withdrawal ameliorates HCV-induced liver damage.

This is a prospective trial in which immunosuppressive drug weaning will be offered to HCV-positive liver recipients (selected on the basis of a high likelihood of tolerance) as a strategy to improve HCV-mediated liver disease.

DETAILED DESCRIPTION:
Objective: To determine the influence of hepatitis C virus (HCV)-driven immune responses on the acquisition of operational tolerance in liver transplant recipients following drug weaning, and to assess whether immunosuppression withdrawal ameliorates HCV-induced liver damage.

Background: Viral infections can profoundly influence alloimmune responses and hamper allograft tolerance induction. Persistent HCV infection occurs in 50% of liver and 20% of kidney transplant recipients, but the impact of HCV on the acquisition of allograft tolerance has not been elucidated. Liver transplantation constitutes a unique clinical model to address this question, given that up to 20% of liver recipients can completely discontinue immunosuppressive drugs and attain operational tolerance.

Hypothesis/Specific Aims: We hypothesize that HCV positive patients failing to attain operational tolerance will exhibit both decreased anti-HCV specific T cell responses and exacerbated non-specific immunoactivation. Furthermore, we anticipate that successful immunosuppression withdrawal will decrease the progression of HCV-induced liver damage. Thus our aims are:

1. To test whether the magnitude of HCV-mediated inflammatory responses influence the acquisition of operational tolerance following liver transplantation.
2. To establish the impact of anti-HCV specific CD4+ and CD8+ T cell immune responses on the capacity of liver recipients to successfully withdraw immunosuppression.
3. To determine how the immunophenotypic traits and functional properties of T cells, NK cells and antigen presenting cells affect the development of operational tolerance in HCV-positive liver recipients.
4. To assess the effect of immunosuppression weaning on the histological progression of HCV-induced liver damage.

Proposed methods: On the basis of a previously identified immunophenotypic signature of tolerance (high ratio of delta 1 to delta 2 gammadelta T cell in peripheral blood), drug weaning will be offered to HCV-positive liver recipients as a strategy to improve HCV-mediated liver disease. We estimate that patients selected on the basis of this biomarker will have a likelihood of successful weaning greater than 50%. Both peripheral blood and liver tissue samples will be collected for diagnostic purposes before the initiation of drug weaning in order to perform the following assays: measurement of anti-HCV CD4+ and CD8+ T cell immunity, peripheral blood and liver tissue gene expression profiling, peripheral blood cell phenotyping and functional assays and, in a subset of patients, measurement of anti-donor T cell responses. Immunosuppression drugs will be weaned over a period of 6 months, and thereafter patients will be followed for 12 additional months. Patients not undergoing rejection during this 18 month period will be considered tolerant. Liver biopsies will be obtained before the beginning of the study and at the end. Progression of HCV-induced liver diseased will be compared to that of patients with a low delta1/delta2 ratio, in whom no changes in immunosuppressive drugs will be conducted and liver biopsies will be obtained yearly (according to our clinical guidelines).

Expected results: We expect to precisely define how HCV influences the acquisition of operational tolerance after liver transplantation, and confirm the beneficial effect of immunosuppression withdrawal in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation for HCV-related liver disease performed at least 3 years before weaning;
* Peripheral blood Vgd1+/Vgd2+ T cell ratio >2.33 and/or increased expression of KLRF1 and SLAMF7 genes in peripheral blood (measured by qPCR).
* No indication for treatment with pegylated a-interferon plus ribavirin during the weaning procedure;
* Stability of liver function tests for at least 6 months;
* No evidences of autoimmune liver disease;
* Absence of acute and/or chronic rejection episodes during the 12 months before weaning;
* Basal liver biopsy without signs of acute and/or chronic rejection.
* Absence of decompensated chronic liver disease.

Exclusion Criteria:

* HIV infection
* Double liver-kidney transplantation
* HCV cholestatic fibrosing hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Proportion of hepatitis C virus positive liver recipients successfully withdrawing immunosuppressive drugs. | 18 months

SECONDARY OUTCOMES:
Effects of immunosuppression withdrawal on hepatitis C virus induced liver damage. | 18 months
Influence of HCV-induced immune responses on the feasibility of successfully withdrawing immunosuppressive drugs in liver transplant recipients. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sanchez-Fueyo, MD, Principal Investigator — Hospital Clinic Barcelona / IDIBAPS, Barcelona, Spain; Giuseppe Tisone, MD, Study Chair — University Tor Vergata, Rome, Italy; Marina Berenguer, MD, Study Chair — Hospital La Fe de Valencia
Locations (1):
- Hospital Clinic Barcelona, University of Barcelona, Barcelona, Spain